CLINICAL TRIAL: NCT02367950
Title: Feasibility and Acceptability of Exercise as a Lifestyle Intervention in Endometrial Cancer Survivors.
Brief Title: Exercise as an Intervention in Endometrial Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Principal Investigator, Khadra Galaal, Consultant Gynaecological Oncologist, Royal Cornwall Hospitals Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014.RCHT.62
Record Dates: First submitted 2015-02-02; First posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Endometrial Cancer; Quality of Life
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Study (Experimental): All participants receive active treatment (exercise) tailored to their level of health ad fitness
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 10 exercise sessions with a personal trainer

SUMMARY:
The purpose of the study is to evaluate the feasibility of introducing an exercise programme for endometrial cancer survivors.

DETAILED DESCRIPTION:
Objectives

* To evaluate the feasibility of an exercise intervention for endometrial cancer survivors in terms of recruitment, adherence, response rates, and follow-up rate.
* To evaluate the feasibility of the individual components of the exercise programme itself within the study population.
* To evaluate if the outcomes measure used to evaluate quality of life outcomes such as psychological distress, fatigue and pain in endometrial cancer survivors are appropriate.
* To evaluate if the outcome measures used to evaluate physical fitness are appropriate.
* To evaluate the acceptability of an exercise intervention for endometrial cancer survivors to improve quality of life outcomes.

General research design Single-arm prospective feasibility study In addition we will conduct a qualitative evaluation with a purposively selected subgroup with maximum variation of our population.

Study population All women diagnosed at the Royal Cornwall Hospital with endometrial cancer who have completed surgical treatment.

Number of participants Every year approximately 90 women are diagnosed with endometrial cancer at the Royal Cornwall Hospital in Truro, of which approximately 80 women receive primary surgical treatment. We estimate that 50% to 60% will consent to participation in this study; we therefore anticipate that the sample size for a study duration of 12 months will be approximately 40 to 48 women.

As this is a feasibility study, we have not performed a power analysis.

Setting Single centre study at the Royal Cornwall Hospital, Truro.

Selection and identification Women with a confirmed diagnosis of endometrial cancer will be introduced to the study by a member of the clinical team post-operatively during admission for surgery.

Identification of potential participants will be performed by a member of the clinical care team (consisting of three gynaecological oncologists, a Clinical Nurse Specialist (CNS) and a clinical research fellow). This will be performed through the review of medical records using case notes and an electronic clinical database system (MAXIMS), before the start of the gynaecological oncologist clinic and during multidisciplinary gynaecological oncology team meetings.

Recruitment Potential participants will be introduced to the study by the clinical care team during their admission for surgical treatment and a study information sheet will be given. Potential participants will be asked if a member of the clinical team can contact them by telephone, one week after they are discharged home, to discuss the study in detail and their possible participation. Following this telephone call, only women who express an interest in participating in the study will be further approached at their next outpatient clinic appointment (6 weeks post-operative). Informed consent for the study will be sought during this patient's clinical visit, which occurs at approximately 6 weeks after the operation. During this process the gynaecological oncologist, the CNS or the clinical research fellow will explain the details of the study, the risks, burdens and possible benefits, and answer any additional questions the patient may have.

Intervention In this study, the intervention itself will be delivered by a male Cancer Exercise Specialist, funded by a local charity 'Active Pants', who provide a post-treatment rehabilitation programme for cancer patients. The programme objectives are to improve health status and promote a healthy lifestyle, and are based on specific and national guidelines (27-29).

Prior to starting the programme, participants receive a health and physical fitness assessment by the Cancer Exercise Specialist. The health assessment will include their current health and physical activity level according to the patient, any medical conditions and medical history, and other restrictions the patient may experience in terms of exercising. The physical fitness assessment will include measuring weight and height, waist circumference, body fat percentage, muscle percentage and resting metabolism and the 6-minute walk test. In addition, any personal goals of the patient will be identified. This will take approximately 30 minutes.

The exercise programme consists of 60-min individualised (one-on-one) personal training sessions, once a week, for 10 weeks. Each session consists of a 10 min warm-up, a 40-min work out, consisting of cardiovascular exercise, pillar strength exercise (including hip and core stability), and resistance training (muscular strength and endurance training), and a 10-min cooling down including flexibility training (see Appendix 3). The programme will be tailored to the individual patient by the Cancer Exercise Specialist, taking into consideration their current health status, comorbidities and medical history. A personal Cancer Exercise Specialist with experience in various cancer areas will supervise the exercise programme one on one with the participant, giving them a specific set of exercised each session, tailored to the individual patient.

After completion of the 10-week supervised exercise programme, participants are given the opportunity to continue their training in weekly group sessions for free, supervised by the same Exercise Specialist.

The Exercise Specialist will document the attendance rates of participants and if participants completed their 10 exercise sessions. The 6-min walk test will be performed after completion of the 10th session of the programme to assess a possible change in physical fitness compared to baseline physical fitness. In addition the Exercise Specialist will document the individual response of participants to components of the exercise sessions and how they were tolerated.

Follow-up Follow-up will take place after completion of the exercise sessions at the standard clinical visit with the gynaecological oncology team, which is 3 to 4 months after the post-operative (6 week) visit. Patients will then come back again after 3 months.

Data management Data will be collected by the clinical care team (gynaecological oncologists, the CNS, and clinical research fellow) when the patients attend for their routine outpatient appointments. The data will be anonymised prior to being analysed by the clinical research fellow on a password secured NHS computer at the Royal Cornwall Hospital in Truro. Data will remain in a password secured file on this computer and will not be transferred onto another medium or outside the hospital Trust. The manual files including the questionnaires will be stored in a locked office within the Royal Cornwall Hospital.

Project Management The day-to-day management of the study will be undertaken by the Chief Investigator with the support of the Clinical Research Fellow. The general conduct and progress of the study will be overseen by a Study Management Group (SMG). This group will comprise the chief investigator, the clinical research fellow and the study data analyst, with occasional attendance by a sponsor's representative and patient representative as required. The SMG will meet often during the study set-up and less frequently once the study is underway with minutes circulated to all SMG members.

The sponsor, Royal Cornwall Hospital, has arrangements in place to monitor or audit the conduct of the study as part of the sponsor's obligations under the Department of Health's Research Governance Framework. The purpose of an audit or inspection is to systematically and independently examine all study related activities and documents to determine whether these activities were conducted, and data were recorded, analysed, and accurately reported according to the protocol, Good Clinical Practice (GCP), ICH guidelines, and any applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of endometrial cancer
* Completion of surgical treatment for endometrial cancer
* Age; 18 years or older.

Exclusion Criteria:

* Women receiving treatment in the palliative setting
* Women with recurrent diagnosis of endometrial cancer
* Women with concurrent cancer
* Women who are unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The number of invited participants that complete the tailored exercise programme (10 exercise sessions). | 18 months
  The overall aim of this proposed feasibility study is to ensure that a larger trial can successfully be planned and delivered.

SECONDARY OUTCOMES:
Change from baseline in the EORCT QLQ-C30 quality of life outcome measures at 18 months and change from baseline in the QLQ-EN24 quality of life outcome measures at 18 months. | 18 months
  The perceived psychological benefits (anxiety and depression) of undertaking physical exercise.
Change from baseline in the Brief Fatigue Inventory outcome measures at 18 months and change from baseline in the Brief Pain Inventory outcome measures at 18 months. | 18 months
  The perceived psychological benefits (fatigue and pain) of undertaking physical exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Cannaby, BA, Study Director — United Kindom: Royal Cornwall Hospital
Locations (1):
- Royal Cornwall Hospital Trust, Truro, Cornwall, United Kingdom

REFERENCES:
- [Derived] Smits A, Lopes A, Das N, Bekkers R, Massuger L, Galaal K. Exercise Programme in Endometrial Cancer; Protocol of the Feasibility and Acceptability Survivorship Trial (EPEC-FAST). BMJ Open. 2015 Dec 16;5(12):e009291. doi: 10.1136/bmjopen-2015-009291. PMID 26674498